CLINICAL TRIAL: NCT01826825
Title: Preoperative Cognitive Screening of Elderly Surgical Patients
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Principal Investigator, Gregory J. Crosby, M.D., Physician, Brigham and Women's Hospital
Other Study IDs: Culley_01
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Impairment
Keywords: aging; cognition; surgery
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clock in the box: Those patients with and without probable cognitive impairment based on the Clock-in-the-box assessment.
  Interventions: Behavioral: Cognitive Screen
- Mini-Cog: Those patients with and without probable cognitive impairment based on the Mini-Cog assessment.
  Interventions: Behavioral: Mini-Cog

INTERVENTIONS:
Behavioral: Cognitive Screen — Cognitive Screen
  Other Names: Clock-in-the-Box
  Groups: Clock in the box
Behavioral: Mini-Cog — Cognitive Screen
  Other Names: Mini-Cog cognitive screen
  Groups: Mini-Cog

SUMMARY:
The objectives of this pilot study are:

1. to determine whether a short cognitive test battery administered in the preadmission test center can be used to cognitively stratify elderly patients presenting for elective surgical procedures.
2. to evaluate the cost of cognitive screening in the preoperative testing center in terms of time and finances.
3. to evaluate patient perceptions about the use of preoperative cognitive screening and their outcome expectations from their surgical procedure.

Subsequent investigations may evaluate whether preoperative cognitive screening is a predictor of postoperative morbidity and mortality in elderly surgical patients and whether a short cognitive screen administered in the preadmission testing center could be used to identify individuals with baseline cognitive impairments that should be refered for more formal cognitive evaluation.

DETAILED DESCRIPTION:
Detailed Description: Background and Significance: Approximately one-third of elective surgical patients seen in the BWH Preoperative Test Center are 65 years of age or older and national trends are similar. 15-30% of community dwelling elders have cognitive impairment. Such impairment cannot be identified based on chronologic age alone because there is considerable heterogeneity in cognitive abilities within and between age groups. In clinical practice, however, the brain is one major organ system that is not assessed formally preoperatively, so those with pre-existing cognitive deficits often go unrecognized. This is a potentially important deficiency given the advanced age of many surgical patients, the difficulty cognitive impairment may impose on ability to follow postoperative instructions, and the fact that research studies show an association between pre-existing cognitive impairment and risk for perioperative morbidity and mortality. Thus, preoperative cognitive performance may be a predictor and/or modifier of postoperative outcomes.1,2,3 Interestingly, no studies have documented patient perceptions regarding relationships between cognitive performance and patient outcomes among elders presenting for elective surgical procedures.

Objectives:

Objective 1: To determine whether each of two short cognitive tests administered in the preadmission test center are equally useful in cognitively stratify elderly patients presenting for elective surgical procedures.

Objective 2: To evaluate the cost of cognitive screening in the preoperative testing center in terms of time and finances.

Objective 3:To evaluate patient perceptions about the use of preoperative cognitive screening and their outcome expectations from their surgical procedure.

Subsequent investigations may evaluate whether preoperative cognitive screening is a predictor of postoperative morbidity and mortality in elderly surgical patients.

Subject Selection: Two hundred patients over age 65 years scheduled for an elective surgical procedure without a planned postoperative admission to the ICU will be identified by the Weiner Center for Preoperative Evaluation (PATC). The study will include patients of both genders scheduled for surgery without planned admission to an ICU. Exclusion criteria include a formal diagnosis of dementia (e.g. Alzheimer's disease), uncorrected vision or hearing impairment (as it is necessary to see pictures and hear instructions), inability to speak, read or understand English, and scheduled surgical procedures affecting the brain or cerebrovasculature (i.e. intracranial neurosurgery, carotid endarterectomy). These ages are chosen because cognitive impairment becomes more prevalent after age 65 years of age and patients in this age group are at greatest risk for developing serious postoperative complications.

Subject Enrollment: The Brigham and Women's Hospital is the only study site. When the patients check in for their preoperative evaluation they will be asked by the registration desk whether a study investigator can discuss the objectives and risks of a study that is being performed in the preadmission testing center. If the patient agrees a member of the investigative team will greet the patient and describe the purpose of study to them along with its risk and benefits and provide them with the consent form for them to read. After the patient has read the consent form they will be asked if they have any additional questions. Once all questions have been answered the patient will be given the opportunity to decline or provide written informed consent to the study.

Study Procedures: After consent is obtained the investigator will thank the patient and open the next available sealed envelop which will contain a study registration ID number and open the envelope wherein the group to which the patient has been randomized will be displayed along with 3 stickers with the registration ID that will be placed on the testing documentation. The Registration ID's will be randomly assigned to a group based on the results of a random number generator.

After randomization the investigator will hand the patient the Patient Survey (see Patient Survey attached) on a clipboard with a pen attached and the patient will compete the survey in the waiting room of the preadmission testing center. Once completed the investigator will collect the survey. If the patient has been randomized to the Clock-in-the-box test they will be handed the instructions to the test and be allowed to read them. After the patient has read the instructions the patient will hand the instructions to the investigator who will place a copy of the test form on the clipboard for the patients use. After the patient has completed the clock-in-a-box test they will return it to the investigator who will thank the patient for their participation in the study. A trained member of the investigative team will score the clock-in-a-box test after the preadmission test center visit. (See attachment A for the Clock-in-the-Box test and scoring).

For patients randomized to the Mini-Cog, a trained member of the preadmission test center team who is involved in the patients routine preoperative evaluation will administer the test during the course of the patients preoperative evaluation in a quiet room. They will first instruct the patient to remember 3 unrelated words (egg, apple, table, penny). The patient will be requested to repeat the words back to the clinician to ensure they heard the words. Next the patient is instructed to draw the face of a clock with the hands on a specific time (the time 11:10 has been endorsed). Finally the patient is instructed to recall the 3 words. The Mini-Cog is scored by giving 1 point for each word recalled, a normal clock is scored as 2 points and an abnormal clock receives 0 points. Mini-Cog scores can range from 0 (worst score) to 5 (best score). Because these studies are not intended to detect dementia nor impact current medical care the test scores will not be released to the patient nor will there be a referral to a neurologist for more formal cognitive evaluation although subsequent investigations may study the value of doing so (see Attachment 2 for Mini-Cog test and scoring).

Other data to be collected will include the age of the patient, the total duration of time the patient spent in the preadmission test center (check-in time to departure time), the duration of their preoperative evaluation (time in the preoperative evaluation room) as identified by the CPE tracking system and the monetary cost of this time in each area and compared to those variables in patients over age 65 presenting for preoperative evaluation the week before and the week after the study period and compared using a Student's t-test.

Biostatistical Analysis: For the Clock-in-the-Box test the number of patients with scores of 0-8 between the ages of 65-74 vs 75 and above will be determined and analyzed using a chi square analysis. For the Mini-Cog test the number of patients with scores of 0-5 for ages 65-74 vs 75 and above will be determined and analyzed using a chi square analysis to determine whether this tool can be used for cognitive stratification in patients in the preadmission testing center. One would expect that older patients would score lower on this test when compared to younger patients.

This study does not involve a medical intervention or treatment or diagnosis of a disease process but rather will determine whether cognitive stratification of elders is feasible within the established flow of the preoperative testing center process of the Brigham and Women's Hospital, the cost of such testing, and patient perceptions regarding the value.

Survey data will be presented as the percentage of patients agreeing with each statement when binary and will provide valuable patient centered insight about their perceptions of preoperative cognitive stratification and their outcome goals resulting from their upcoming surgical procedure.

Data on duration of time spent in the preadmission testing center and duration of 1:1 preoperative evaluation for study versus non-study patients over the age of 65 will be analyzed using a Student's t-test.

Risks and Discomforts:

Risks to patients are minimal, as the cognitive screening results will only be reported in aggregate with no personally identifiable information. The cognitive screen will have no impact on patient care and thus should not alter patient outcomes although some patients may experience stress if they are having difficulty with the cognitive exam. All efforts will be made to minimize risks by selecting investigators who are trained to the protocol and cued to monitor the patient for undo stress. Patient participation in the study can be discontinued at any time if the opinion of the investigator is that it is in the best interest of the patient to discontinue participation or if the patient requests withdrawal from the study

Potential Benefits:

There are no expected benefits to individual subjects participating in the study. This study has the potential to aid and improve decision-making by physicians and elderly patients in the future if they reveal a relationship between poor preoperative cognitive status and adverse postoperative outcomes in elders.

Monitoring and Quality Assurance:

Regardless of monitoring plans, the principal investigator is ultimately responsible for ensuring that the study is conducted at his/her investigative site in accordance with the IRB-approved protocol and applicable regulations and requirements of the IRB.

The Principal Investigator or a member of the investigative team will monitor each subject at this single site, and will review the accuracy and completeness of Clock-in the Box, Mini-cog and survey reports, source documents and informed consent.

There will be no Data Safety Monitoring Board as the results of these studies will have no impact on the care that patients receive. The outcomes of the study are intended to be published in a peer-reviewed manuscript. All adverse events will be reported to the Partners the Human Research Committee (HRC) in accordance HRC guidelines. A 24-hour/7-day telephone or pager number will be provided for contacting the licensed physician investigator for this purpose.

The research staff will monitor all subjects during the course of study involvement for evidence of any adverse events such as unexpected stress and the testing discontinued and the incident reported to Partners the Human Research Committee within 24 hours of local event awareness (but no later than the next business day). The report will include a complete description of the event, use of all concomitant medications, and the local investigator's assessment of causality of the adverse event. Follow-up evaluations will be done until there is resolution of the adverse events, which are unlikely as this protocol is non-invasive

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years and over were enrolled either to be screened with the Clock in the Box or MiniCog cognitive screening tools

Exclusion Criteria:.

* Patients under age 65 Patients with visual or hearing impairments that are not corrected Patients who do not speak and read English Patients having a formal diagnosis of dementia Patients with scheduled surgical procedures affecting the brain or cerebrovasculature (i.e. intracranial neurosurgery, carotid endarterectomy).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 200 patients over the age of 65 that have provided informed consent will be randomly assigned to either the mini-cog or the clock in the box cognitive screen.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bader, MD, MPH, Study Chair — Brigham and Women's Hospital; James Rudolph, MD, Study Chair — Brigham Hospital; Deborah J Culley, MD, Principal Investigator — Brigham Hospital; Devon M Flaherty, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the Preadmission Testing Center at BWH between 6/5/2013 and 7/31/2013 after completing the informed consent process.
Pre-assignment Details: 2 patients initially agreed to participate in the study but then were called in for their preadmission appointment and were not enrolled.
Groups:
- Clock in the Box: Results of the Clock in the box cognitive screening test.
  Cognitive Screen: Cognitive Screen
- Mini-Cog: Results of the mini-cog cognitive screen
  Mini-Cog: Cognitive Screen
Period: Overall Study
Arm/Group | Clock in the Box | Mini-Cog
Started | 100 | 100
Completed | 100 | 98
Not Completed | 0 | 2
Not completed — Two patients consented and randomized to Mini-Cog did not have the Mini-Cog administered | 0 | 2

BASELINE CHARACTERISTICS:
Population: 2 Patients enrolled in the Mini-Cog group withdrew from the study before MiniCog administration
Groups:
- Total: Total of all reporting groups
Arm/Group | Clock in the Box | Mini-Cog | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants] — All patients enrolled were 65 years of age and older
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 100 | 100 | 200
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 Patients withdrew
  Participants
    number analyzed (Participants) | 100 | 98 | 198
    Female | 50 | 50 | 100
    Male | 50 | 48 | 98
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Probable Cognitive Impairment
Description: Potential baseline predictors of the MiniCog and CIB scores on a risk ratio scale, Clock in box 0-8, Mini-Cog 0-5, higher values represent better scores. For the Mini-cog a score of less than or equal to 2 suggests probable cognitive impairment. For the Clock in the box, a score of less than or equal to 5 suggests probable cognitive impairment. The number of participants that scored less than or equal to 2 on the Mini-cog or less than or equal to 5 on the clock in the box are presented in the data table
Time Frame: Cognitive stratification occurred on the date the patient consented to the study at baseline. This data was presented in a publication in 2017 (Anesthesiology. 2017 Nov;127(5):765-774.)
Population: Mini-Cog less than or equal to 2, clock in the box scores less than or equal to 5 suggests probable cognitive impairment
Measure: Count of Participants; unit: Participants
Arm/Group | Clock in the Box | Mini-Cog
Number analyzed (Participants) | 100 | 98
Participants | 23 | 22

2. Secondary Outcome: Cost of Cognitive Screening in Terms of Time and Finances
Description: To evaluate the cost of cognitive screening in the preoperative testing center in terms of time and finances. We were unable to determine differences in cost and did not track time to administer specifically the screening tools but rather the time of the entire preoperative evaluation. We gathered information on time spent in the preoperative testing center between patients who had MiniCog or Clock-in-the box testing.
Time Frame: duration of time undergoing preoperative evaluation in minutes.
Population: Study patients undergoing cognitive screening with either the MiniCog or Clock in the Box.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- MiniCog: Duration of the preoperative evaluation for patients randomized to the MiniCog cognitive screen.
- Clock in the Box: Duration of the preoperative evaluation for patients randomized to the Clock in the Box cognitive screen.
Arm/Group | MiniCog | Clock in the Box
Number analyzed (Participants) | 82 | 84
Minutes | 90 (38) | 90 (38)

3. Secondary Outcome: Patient Perceptions of Preoperative Cognitive Screening
Description: Results of a patient survey about their perceptions on preoperative cognitive screening on a yes / no basis
Time Frame: The data was obtained at the time of initial enrollment
Population: Patient perspective of preoperative cognitive screening. Because 2 patients randomized to the MIni-Cog arm were taken in for their preoperative assessment neither the Mini-cog screen and the survey on their perceptions on preoperative cognitive screening were obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Clock in the Box | Mini-Cog
Number analyzed (Participants) | 100 | 98
Participants
  Do you believe a short memory test should be performed before having a surgical procedure?: Yes | 71 | 71
  Do you believe a short memory test should be performed before having a surgical procedure?: No | 19 | 9
  Do you believe a short memory test should be performed before having a surgical procedure?: Refused to answer | 10 | 18
  If a memory test could help predict surgical outcomes would you want memory testing performed?: Yes | 92 | 93
  If a memory test could help predict surgical outcomes would you want memory testing performed?: No | 3 | 3
  If a memory test could help predict surgical outcomes would you want memory testing performed?: Refused to answer | 5 | 2
  If the results of memory testing suggested memory problems would you want to know?: Yes | 93 | 93
  If the results of memory testing suggested memory problems would you want to know?: No | 5 | 5
  If the results of memory testing suggested memory problems would you want to know?: Refused to answer | 2 | 0
  If the memory test suggested possible memory problems would you want a memory specialist referral?: Yes | 80 | 75
  If the memory test suggested possible memory problems would you want a memory specialist referral?: No | 15 | 20
  If the memory test suggested possible memory problems would you want a memory specialist referral?: Refused to answer | 5 | 3

ADVERSE EVENTS:
Time Frame: In hospital, and up to 1 month postoperatively. This data was collected from the patients chart between 1 month and 2 months after their surgical procedure.
Arm/Group | Clock in the Box | Mini-Cog
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/98
Serious Adverse Events (participants affected / at risk) | 13/100 | 18/98
Other Adverse Events (participants affected / at risk) | 0/100 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clock in the Box (N=100) | Mini-Cog (N=98)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Postoperative pneumonia
Reintubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient reintubated during their hospital stay
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — In hospital postoperative stroke
Delirium by Chart review (Nervous system disorders) | 7 (7) | 8 (8) — In hospital delirium by chart review
Wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — In hospital wound infection
Sepsis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — In hospital postoperative sepsis
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 3 (3) — Postoperative urinary tract infection
Reoperation (Surgical and medical procedures) | 2 (2) | 4 (4) — Reoperation during hospitalization in the postoperative period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes